CLINICAL TRIAL: NCT01775254
Title: Self Reported Changes in Quality of Life, Demands of Illness, and Sexual Function in Colon Cancer Survivors.
Brief Title: The Inland Northwest Colon Cancer Survivor's Study
Status: Completed | Type: Observational
Sponsor: Washington State University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: DSCN-11-194-01
Record Dates: First submitted 2013-01-23; First posted 2013-01-24 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Colon Cancer
Keywords: Colon Cancer; FOLFOX; Laparoscopic Colectomy; Open Colectomy; Robotic Colectomy; Quality of Life; Sexual Function; Peripheral Neuropathy; Demands of Illness; Cancer Survivor
MeSH Terms: conditions — Colonic Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chemotherapy Group: Colon cancer survivors who undergo open or laparoscopic resection of their colon cancers followed by adjuvant chemotherapy.
- No Chemotherapy Group: Colon cancer survivors who undergo open or laparoscopic resection of their colon cancer and who do not receive chemotherapy.

SUMMARY:
The overall purpose of this study was to address the following questions by describing the trajectory of early survivorship in individuals who undergo both surgical and medical management of colon cancer. What are the changes in quality of life, demands of illness, sexual function, and peripheral neuropathy, following curative resection during the first year of treatment and recovery? Is there an interaction between exposures to chemotherapy and changes over time in these outcomes?

DETAILED DESCRIPTION:
The population of interest included colon cancer survivors of both sexes, 18 to 90 years of age, who underwent one of two types of surgical resection and who may receive adjuvant chemotherapy. The prospective design with two cohorts representing exposure to chemotherapy (chemotherapy vs. no-chemotherapy) described the changes in quality of life, demands of illness, sexual function, and peripheral neuropathy, which occurred following curative resection. An analysis of the interaction between time (four measurement occasions) and the independent variable of chemotherapy group by mean values of quality of life, sexual function, peripheral neuropathy, and demands of illness addressed the central thesis question.

Specific Aims

1. Examine the relationships among quality of life, demands of illness, sexual functioning, and peripheral neuropathy, for the total sample and by chemotherapy group.
2. Examine changes within-subjects (four measurement occasions), between-group (chemotherapy, no-chemotherapy) differences, and the interaction between time and chemotherapy group for quality of life, demands of illness, sexual functioning, and peripheral neuropathy across four measurement occasions.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age
* Biopsy Proven Colon Cancer
* Plan to undergo open, laparoscopic or robotic surgical colectomy.

Exclusion Criteria:

* Persons with rectal cancer
* Surgical resection below the rectal sigmoid junction
* Does not speak or read English
* Scheduled to receive radiation therapy during the data collection period
* Diagnosis of metastatic colon cancer (Stage IV)
* A previous history of cancer diagnosed with the past five years with the exception of early basal cell or squamous skin cancer or early stage melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons newly diagnosed with colon cancer anticipated to undergo curative resection. To include those who will receive adjuvant FOLFOX chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10-15 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Four measurements occasions over 42 weeks (Before surgery, 4-6 weeks after surgery, 20-24 weeks after surgery and 32-36 weeks after surgery)
  The European Organization for Research and Treatment Quality of Life Questionnaire

SECONDARY OUTCOMES:
Change in Peripheral Neuropathy | Four measurements occasions over 42 weeks (Before surgery, 4-6 weeks after surgery, 20-24 weeks after surgery and 32-36 weeks after surgery)
  The Neurotoxicity Sub-scale (Ntx-13); a questionnaire about symptoms of nerve damage in persons receiving chemotherapy, will be utilized to assess symptoms of neurologic toxicities in persons receiving the chemotherapy drug oxaliplatin. The interaction between time (four measurement occasions) and chemotherapy group (chemotherapy, no chemotherapy ) by mean values of peripheral neuropathy will be examined.
Change in Sexual Function | Four measurements occasions over 42 weeks (Before surgery, 4-6 weeks after surgery, 20-24 weeks after surgery and 32-36 weeks after surgery)
  Change in Sexual Function Questionnaire (CSFQ)will be used to describe the changes in sexual function reported by cancer survivors following surgery and adjuvant chemotherapy. The interaction between time (four measurement occasions) and chemotherapy group (chemotherapy, no chemotherapy ) by mean values of changes in sexual function will be examined.
Change in Patient Education and Support Utilized | Four measurements occasions over 42 weeks (Before surgery, 4-6 weeks after surgery, 20-24 weeks after surgery and 32-36 weeks after surgery)
  A short questionnaire regarding the use of educational and support materials related to colon cancer will be used to describe which materials persons with colon cancer utilize during the 8 months after diagnosis.
Change in Demands of Illness | Four measurements occasions over 42 weeks (Before surgery, 4-6 weeks after surgery, 20-24 weeks after surgery and 32-36 weeks after surgery)
  The Demands of Illness Inventory (DOII); a questionnaire about the stressors experienced by cancer survivors will be utilized for this outcome measure. The interaction between time (four measurement occasions) and chemotherapy group (chemotherapy, no chemotherapy ) by mean values from the demands of illness inventory will be examined.

OTHER OUTCOMES:
Psychometric analysis of a modified version of the Neurotoxicity Sub-scale. | At the completion of the study
  Psychometric analysis to evaluate the reliability and validity of the modified Neurotoxicity Sub-Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Robison, PhD, ARNP, Principal Investigator — Washington State University, College of Nursing; Mel Haberman, PhD, FAAN, Principal Investigator — Washington State University, College of Nursing
Locations (4):
- United States (4):
  - Deaconess Hospital, Spokane, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - Holy Family Hospital, Spokane, Washington
  - Valley Hospital, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No